CLINICAL TRIAL: NCT07060352
Title: Estimating the Prevalence of GAstrocnemius Muscle REtraction in a Population Suffering From Plantar aPOneurositis and Describing the Effects of Lengthening
Acronym: REGAPOP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Charles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REGAPOP; 2025-A00798-41 (Other: ANSM)
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ankle Dorsiflexion Index (ADI) measurement (Experimental): Ankle Dorsiflexion Index (ADI) measurement at D0 and W8
  Interventions: Diagnostic Test: Ankle Dorsiflexion Index (ADI) measurement

INTERVENTIONS:
Diagnostic Test: Ankle Dorsiflexion Index (ADI) measurement — Ankle Dorsiflexion Index (ADI) measurement at D0 and W8

SUMMARY:
The gastrocnemius muscles, which form the upper part of the calf, can suffer from retraction, a common but often under-diagnosed condition, which can be a risk factor for plantar fasciitis. Retraction can be treated medically, by stretching, or surgically, by lengthening the muscles. Gastrocnemius retraction is difficult to measure, but tests such as the Ankle Dorsiflexion Index (ADI) provide a more accurate assessment.

Knowing the prevalence of this retraction in patients suffering from plantar fasciitis would enable us to improve diagnostic criteria and better target treatments. Surgical lengthening of the gastrocnemius, particularly by tenotomy, is effective in cases of chronic plantar fasciitis, even without apparent muscle retraction.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 70 or under
* Patient suffering from unilateral plantar fasciitis that has progressed for more than 6 months and is recalcitrant to medical treatment
* Collection of express, oral consent
* Available for follow-up visits

Exclusion Criteria:

* Patients with neuropathic pain
* History of fracture of the lower limb, surgery on the lower limb, inflammatory rheumatism of the lower limb, injury to the Achilles tendon
* Patient with another painful orthopedic lesion of the legs/feet
* Patient with surgically treated plantar fasciitis in the year prior to inclusion
* Persons unable to give consent
* Not affiliated to a social security scheme
* Persons under court protection
* Participant in another study with an ongoing exclusion period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gastrocnemius muscle retraction in patients with plantar fasciitis | At Day 0
  retraction of the gastrocnemius muscles will be defined by an ADI of less than 13° measured by a digital inclinometer

SECONDARY OUTCOMES:
correlation between ADI measurement and Manchester Oxford Foot Questionnaire (MOXFQ) | At Day 0
  The Manchester Oxford Foot Questionnaire (MOXFQ) is used to measure the impact of foot pain on patients' quality of life. It consists of 16 questions. The raw scores of the scales are converted into a metric scale ranging from 0 to 100, where 100 indicates the maximum intensity of suffering or limitation.
correlation between ADI measurement and pain Visual Analog Scale (VAS) | At Day 0
  The VAS consists of a straight line where one extreme represents the total absence of pain and the other extreme, the most intense pain possible. Patients are asked to mark on this line the level of pain they feel at any given moment. Pain intensity is then measured according to the distance between the start of the scale (0) and the point where the patient placed his mark:
  * 0 cm (or the start of the scale): No pain
  * 10 cm (or the end of the scale): Maximum imaginable pain
Evolution of Visual Analog Scale (VAS) | between Day 0 and Week 8
  The VAS consists of a straight line where one extreme represents the total absence of pain and the other extreme, the most intense pain possible. Patients are asked to mark on this line the level of pain they feel at any given moment. Pain intensity is then measured according to the distance between the start of the scale (0) and the point where the patient placed his mark: - 0 cm (or the start of the scale): No pain - 10 cm (or the end of the scale): Maximum imaginable pain
Evolution of Visual Analog Scale (VAS) | between Day 0 and Week 16
  The VAS consists of a straight line where one extreme represents the total absence of pain and the other extreme, the most intense pain possible. Patients are asked to mark on this line the level of pain they feel at any given moment. Pain intensity is then measured according to the distance between the start of the scale (0) and the point where the patient placed his mark: - 0 cm (or the start of the scale): No pain - 10 cm (or the end of the scale): Maximum imaginable pain
Evolution of Visual Analog Scale (VAS) | between Day0 and Week 24
  The VAS consists of a straight line where one extreme represents the total absence of pain and the other extreme, the most intense pain possible. Patients are asked to mark on this line the level of pain they feel at any given moment. Pain intensity is then measured according to the distance between the start of the scale (0) and the point where the patient placed his mark: - 0 cm (or the start of the scale): No pain - 10 cm (or the end of the scale): Maximum imaginable pain
Evolution of Manchester Oxford Foot Questionnaire (MOXFQ) | between Day 0 and Week 8
  The Manchester Oxford Foot Questionnaire (MOXFQ) is used to measure the impact of foot pain on patients' quality of life. It consists of 16 questions. The raw scores of the scales are converted into a metric scale ranging from 0 to 100, where 100 indicates the maximum intensity of suffering or limitation.
Evolution of Manchester Oxford Foot Questionnaire (MOXFQ) | between Day 0 and Week 16
  The Manchester Oxford Foot Questionnaire (MOXFQ) is used to measure the impact of foot pain on patients' quality of life. It consists of 16 questions. The raw scores of the scales are converted into a metric scale ranging from 0 to 100, where 100 indicates the maximum intensity of suffering or limitation.
Evolution of Manchester Oxford Foot Questionnaire (MOXFQ) | between Day 0 and Week 24
  The Manchester Oxford Foot Questionnaire (MOXFQ) is used to measure the impact of foot pain on patients' quality of life. It consists of 16 questions. The raw scores of the scales are converted into a metric scale ranging from 0 to 100, where 100 indicates the maximum intensity of suffering or limitation.
Correlation between surgical success and body mass index (BMI) | At Day 0
  Surgical success is based on variation of pain (mesured with Visual Analogic Scale)
Correlation between surgical success and age of patient | At Day 0
  Surgical success is based on variation of pain (mesured with Visual Analogic Scale)
Correlation between surgical success and tobacco consumption | At Day 0
  Surgical success is based on variation of pain (mesured with Visual Analogic Scale)
Correlation between surgical success and location of fasciitis | At Day 0
  Surgical success is based on variation of pain (mesured with Visual Analogic Scale) Location of fasciitis: proximal or central

IPD SHARING:
Plan to Share IPD: Undecided